CLINICAL TRIAL: NCT05505331
Title: Three-Dimensional Ultrasonography Versus Magnetic Resonance Imaging for Fibroid Mapping: A Cross Sectional Observational Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Abdelmawgoud, mahmoud abdelMawjud, Sohag University
Other Study IDs: Soh-Med-22-08-02
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Three-Dimensional Ultrasonography Versus Magnetic Resonance Imaging for Fibroid Mapping
Keywords: 3D-Ultrasonography; MRI; Fibroid Mapping
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Uterine Myomectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Radiation: three-Dimensional ultrasonography — transadominal and transvaginal examination
Radiation: Magnetic resonance imaging — multiplanar T2-weighted sequences and pre-contrast T1-weighted imaging in either the sagittal or axial plane
Procedure: myomectomy — myoma excision

SUMMARY:
Three-Dimensional Ultrasonography versus Magnetic Resonance Imaging for Fibroid Mapping: A Cross sectional Observational study

DETAILED DESCRIPTION:
2) Introduction: Uterine fibroids are the most prevalent gynecologic tumors, affecting nearly (20-30) % of women in the reproductive age group[1] . Approximately 50% of fibroid cases are symptomatic [2] and presented by abnormal uterine bleeding, dysmenorrhea, pressure symptoms, infertility, and pregnancy loss[3]. Fibroids are myometrium-derived monoclonal smooth muscle cancers and their growth is reliant on estrogen and progesterone levels, thus fibroids usually expand during pregnancy or during the use of combined oral contraceptives, and shrink after menopause[4]. Two dimensional ultrasound is the initial test of choice to assess the presence of fibroids in symptomatic patients as it is simple, easy, available and informative [5]. Furthermore, ultrasonography may be sufficient for individuals having conservative therapy. However, Magnetic Resonance Imaging (MRI) gives a more precise evaluation of the quantity, location, and type of fibroids specially in cases with considerable uterine enlargement [6, 7] and submucosal fibroids. Furthermore, MRI can be utilized to differentiate between fibroids and their imitators, such as adenomyosis, ovarian neoplasms, and localized myometrial contractions [8].The introduction of 3D ultrasound in evaluating uterine fibroids appears to be an upcoming and promising prospect [9]. However, the evidence on the role of Three-Dimensional Ultrasonography for fibroid mapping is quite limited up till now.

3) Aim of the study The aim of this study is to compare the accuracy of 3D ultrasound and MRI for fibroid mapping in women with symptomatic fibroids diagnosed by 2D ultrasound.

4) Subjects and Methods

1. Study type: Cross sectional observational study
2. Inclusion criteria:

   • Age group: child bearing period.

   • Abnormal uterine bleeding
   * Dysmenorrhea
   * Pressure symptoms
   * Infertility
   * Pregnancy loss
3. Exclusion criteria

   * The cardiac implantable electronic device (CIED)
   * Metallic intraocular foreign bodies
   * Implantable neurostimulation systems
   * Cochlear implants/ear implant
   * Drug infusion pumps
   * Cerebral artery aneurysm clips
   * Magnetic dental implants
   * Artificial limb
4. Methods

   * This study is a clinical trial that will include all patients fulfilling the eligibility criteria and presented to the department of Obstetrics and Gynecology in Sohag University hospital (Egyptian tertiary referral hospital) from August 2022 to July 2023. The attending physician will explain the nature of the study and all patients will be asked to sign an informed consent. All patients underwent gynecologic and ultrasound examinations, comprising standard 2D followed by 3D ultrasound. For both examinations, a transabdominal and transvaginal US (Voluson,p8) will be used. All symptomatic patients who are diagnosed by conventional 2D scan will be subjected to 3D ultrasound in the mid-cyclic period (late follicular phase) and all the following points will be assessed for fibroid mapping.

     o Uterine corpus: Measurement of length, anteroposterior diameter, transverse diameter and volume

     o Serosal contour: Regular versus lobulated

     o Myometrial walls: Symmetrical versus asymmetrical

     o Myometrial echogenicity: Homogeneous versus heterogeneous

     o Myometrial lesions Well defined versus ill defined Number Location (anterior, posterior, fundal, right or left lateral, global) Site (type according to FIGO classification) Size (three perpendicular diameters) Outer lesion-free margin (distance from the serosal surface) Inner lesion-free margin (distance from the endometrial surface) Echogenicity (homogeneous versus heterogeneous; hypo-, iso-, hyper-echogenic)
   * Sonographic evaluation will be done by the same gynecologist to avoid interpersonal variability.

   Then all the patients will be subjected pelvic MRI at the radiology department in Sohag University hospital and all cases will be evaluated by the same radiologist using the proper MRI protocol including multiplanar T2-weighted sequences and pre-contrast T1-weighted imaging in either the sagittal or axial plane. Then we will compare the 3D ultrasonographic evaluation and the MRI fibroid mapping with the definite intraoperative findings and retrospectively evaluate the impact of this evaluation on the selected surgical intervention.
5. Diagnosis of Fibroids by 3D-ultrasonography • This technology captures serial consecutive 2D pictures in three planes: axial, horizontal, and perpendicular. The 2D slice thickness, which may be modified in increments of 2, 4, or 8 mm depending on the individual needs of each investigation, is then translated into volume data, which can subsequently be saved and analyzed in various angles and arbitrary planes[10] . 3D US also offers an accurate coronal view of the uterus, which aids in the delineation of fibroid extension inside the myometrium and into the endometrial cavity. It also depicts the extent and grade of cavity distortion.

3) Outcome measures:

1. Primary

   • The sensitivity and specificity of the 3D-Ultrasonography and MRI for the mapping of different types of symptomatic uterine fibroids according to the final intraoperative diagnosis.
2. Secondary • The validity of 3D-ultrasonography and MRI of Fibroids for selecting the appropriate way of management.

5) Statistical analysis: This is a cross sectional study that will include all eligible patients from August 2022 to July 2023. Case by case analysis will be done to test the sensitivity and specificity of each 3D ultrasonographic marker and MRI for fibroid mapping in comparison to final intraoperative findings. Data will be expressed as mean ± standard deviation (SD), unless stated otherwise. Chi-squared test will be used to compare categorical variables and Student's t-test to compare continuous variables. A p-value of <0.05 will be considered statistically significant. STATA v14 (StataCorp. 2015. Stata Statistical Software: Release 14. College Station, TX: StataCorp LP) and MedCalc programs and will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Age group: child bearing period.

  * Abnormal uterine bleeding
  * Dysmenorrhea
  * Pressure symptoms
  * Infertility
  * Pregnancy loss

Exclusion Criteria:

* • The cardiac implantable electronic device (CIED)

  * Metallic intraocular foreign bodies
  * Implantable neurostimulation systems
  * Cochlear implants/ear implant
  * Drug infusion pumps
  * Cerebral artery aneurysm clips
  * Magnetic dental implants
  * Artificial limb

Ages: 12 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: * Age group: child bearing period.
  * Abnormal uterine bleeding
  * Dysmenorrhea
  * Pressure symptoms
  * Infertility
  * Pregnancy loss
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
• The sensitivity and specificity of the 3D-Ultrasonography and MRI for the mapping of different types of symptomatic uterine fibroids according to the final intraoperative diagnosis | from august 2022 to july 2023
  comparing the ability of 3D-ultrasonography and MRI to detect the exact location of uterine myomas

SECONDARY OUTCOMES:
• The validity of 3D-ultrasonography and MRI of Fibroids for selecting the appropriate way of management | august 2023 to july 2023
  selecting the type of management according to the 3D-ultrasonography as a cheap method

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bulun SE. Uterine fibroids. N Engl J Med. 2013 Oct 3;369(14):1344-55. doi: 10.1056/NEJMra1209993. No abstract available. PMID 24088094
- [Background] McLucas B. Diagnosis, imaging and anatomical classification of uterine fibroids. Best Pract Res Clin Obstet Gynaecol. 2008 Aug;22(4):627-42. doi: 10.1016/j.bpobgyn.2008.01.006. Epub 2008 Mar 7. PMID 18328787
- [Background] Dueholm M, Lundorf E, Hansen ES, Ledertoug S, Olesen F. Accuracy of magnetic resonance imaging and transvaginal ultrasonography in the diagnosis, mapping, and measurement of uterine myomas. Am J Obstet Gynecol. 2002 Mar;186(3):409-15. doi: 10.1067/mob.2002.121725. PMID 11904599
- [Background] Hossain MZ, Rahman MM, Ullah MM, Mukthadira M, Akter FA, Jahan AB, Jahan F. A Comparative Study of Magnetic Resonance Imaging and Transabdominal Ultrasonography for the Diagnosis and Evaluation of Uterine Fibroids. Mymensingh Med J. 2017 Oct;26(4):821-827. PMID 29208870
- [Background] Murase E, Siegelman ES, Outwater EK, Perez-Jaffe LA, Tureck RW. Uterine leiomyomas: histopathologic features, MR imaging findings, differential diagnosis, and treatment. Radiographics. 1999 Sep-Oct;19(5):1179-97. doi: 10.1148/radiographics.19.5.g99se131179. PMID 10489175
- [Background] Saravelos SH, Jayaprakasan K, Ojha K, Li TC. Assessment of the uterus with three-dimensional ultrasound in women undergoing ART. Hum Reprod Update. 2017 Mar 1;23(2):188-210. doi: 10.1093/humupd/dmw040. PMID 28007752
- [Background] Salim R, Lee C, Davies A, Jolaoso B, Ofuasia E, Jurkovic D. A comparative study of three-dimensional saline infusion sonohysterography and diagnostic hysteroscopy for the classification of submucous fibroids. Hum Reprod. 2005 Jan;20(1):253-7. doi: 10.1093/humrep/deh557. Epub 2004 Oct 21. PMID 15498782
- [Result] Deshmukh SP, Gonsalves CF, Guglielmo FF, Mitchell DG. Role of MR imaging of uterine leiomyomas before and after embolization. Radiographics. 2012 Oct;32(6):E251-81. doi: 10.1148/rg.326125517. PMID 23065174
- [Result] Baird DD, Dunson DB, Hill MC, Cousins D, Schectman JM. High cumulative incidence of uterine leiomyoma in black and white women: ultrasound evidence. Am J Obstet Gynecol. 2003 Jan;188(1):100-7. doi: 10.1067/mob.2003.99. PMID 12548202
- [Result] Buttram VC Jr, Reiter RC. Uterine leiomyomata: etiology, symptomatology, and management. Fertil Steril. 1981 Oct;36(4):433-45. doi: 10.1016/s0015-0282(16)45789-4. PMID 7026295